CLINICAL TRIAL: NCT00841789
Title: A Randomized, Double Blind, Placebo Controlled Study of the Effects of Etanercept in Children Presenting With Kawasaki Disease
Brief Title: A Randomized, Double Blind, Placebo Controlled Study of Etanercept in Children With Kawasaki Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Portman (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Michael Portman, Cardiologist, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEA-12652; FD003526 (Other Grant/Funding Number: FD)
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Mucocutaneous Lymph Node Syndrome; Kawasaki Disease
Keywords: Etanercept
MeSH Terms: conditions — Mucocutaneous Lymph Node Syndrome | interventions — Etanercept

STUDY DESIGN:
Intervention Model Description: Approximately 200 subjects will be randomized in a 1:1 ratio to receive Etanercept or Placebo. Subjects are randomized after hospital admission and diagnosis of Kawasaki Disease at eight participating sites. The primary analysis time-point is visit 5 (day 44). Sample size calculation is based on initial IVIG refractory rate at Seattle Children's. Assuming a 17.4% refractory rate in the control group and a 4.3% refractory rate in the Etanercept group, 200 subjects will provide 80% power at a 5% 2-sided type I error rate. Analyses will be based on a modified intention to treat population, including all subjects who were randomized and received at least 1 dose of study drug. Efficacy analyses will be based on randomization assignment, and safety analyses will be based on the treatment actually received. The statistical analysis plan will be finalized prior to database lock and study unblinding.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 -Etanercept (Experimental): Drug - Treatment with Etanercept as adjunct to standard treatment with IVIG and aspirin
  Interventions: Drug: Etanercept
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Etanercept — etanercept 0.8 mg/kg subcutaneously (max 50 mg) given three times, once a week for three weeks starting at initial diagnosis.
  Other Names: Enbrel
  Arms: Arm 1 -Etanercept
Drug: Placebo — Placebo 0.8 mg/kg subcutaneously (max 50 mg) given three times, once a week for three weeks starting at initial diagnosis.
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Etanercept (Enbrel) when used in conjunction with IVIG and aspirin, improves treatment response to IVIG in patients with Kawasaki Disease. Funding Source- FDA/OOPD

DETAILED DESCRIPTION:
Kawasaki Disease (KD) is a potentially life threatening acute vasculitis in children with a predilection for involvement of the coronary arteries. Aspirin and Intravenous gamma globulin (IVIG) are principally used for the treatment of the symptoms of Kawasaki Disease. Aspirin reduces inflammation and platelet formation, but has no effect in attenuating the development of coronary abnormalities. Although IVIG reduces inflammation and the prevalence of coronary artery abnormalities, it has a relatively high failure rate of 23-30%, warranting new treatment methods for Kawasaki Disease. We propose a placebo controlled double blinded randomized study to determine if etanercept 0.8 mg/kg subcutaneously (max 25 mg) given three times at weekly intervals starting at initial diagnosis is safe in this patient population and if it is a successful adjunct therapy with IVIG in reducing the incidence of persistent or recurrent fever.

ELIGIBILITY:
Inclusion Criteria:

* Male Age 2 months to 20 years of age Female Age 2 months to 11 years of age
* Provision of Parental Consent
* Kawasaki Disease Presentation

Exclusion Criteria:

* Laboratory Criteria: Any laboratory toxicity, at the time of the screening visit or at any time during the study that in the opinion of the Investigator would preclude participation in the study or:

  1. Platelet count < 100,000/mm3
  2. WBC count < 3,000 cells/mm3
  3. Hemoglobin, hematocrit, or red blood cell count outside 30% of the upper or lower limits of normal for the Lab
* Subject is currently enrolled in another investigational device or drug trial(s), or subject has received other investigational agent(s) within 28 days of baseline visit.
* Female subjects diagnosed with KD 12 years of age and older.
* Subjects who have known hypersensitivity to Enbrel or any of its components or who is known to have antibodies to etanercept
* Prior or concurrent cyclophosphamide therapy
* Prior treatment with any TNF alpha antagonist or steroid within 48 hours prior to initiation of IVIG
* Concurrent sulfasalazine therapy
* Active severe infections within 4 weeks before screening visit, or between the screening and baseline visits.
* SLE, history of multiple sclerosis, transverse myelitis, optic neuritis, or chronic seizure disorder
* Known HIV-positive status or known history of any other immuno-suppressing disease.
* Any mycobacterial disease or high risk factors for tuberculosis, such as family member with TB or taking INH
* Untreated Lyme disease
* Severe comorbidities (diabetes mellitus requiring insulin, CHF of any severity, MI, CVA or TIA within 3 months of screening visit, unstable angina pectoris, uncontrolled hypertension (sitting systolic BP > 160 or diastolic BP > 100 mm Hg), oxygen-dependent severe pulmonary disease, history of cancer within 5 years [other than resected cutaneous basal or squamous cell carcinoma or in situ cervical cancer])
* Exposure to hepatitis B or hepatitis C or high risk factors such as intravenous drug abuse in patient's mother, or history of jaundice (other than neonatal jaundice). SLE, history of multiple sclerosis, transverse myelitis, optic neuritis or chronic seizure disorder.
* Use of a live vaccine (Measles Mumps Rubella or Varicella) 30 days prior to or during this study.
* Any condition judged by the patient's physician to cause this clinical trial to be detrimental to the patient
* History of non-compliance with other therapies
* Must not have received immunosuppressive agents for at least three months prior to enrollment.

Ages: 2 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 205 (Actual)
Dates: Start 2009-03; Primary Completion 2018-01 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Portman, MD, Principal Investigator — Seattle Children's Hospital
Locations (8):
- United States (7):
  - Feinstein Institute for Medical Rsearch, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Texas Children's Hospital, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Sainte-Justine Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Background] Portman MA, Olson A, Soriano B, Dahdah N, Williams R, Kirkpatrick E. Etanercept as adjunctive treatment for acute Kawasaki disease: study design and rationale. Am Heart J. 2011 Mar;161(3):494-9. doi: 10.1016/j.ahj.2010.12.003. PMID 21392603
- [Result] Portman MA, Dahdah NS, Slee A, Olson AK, Choueiter NF, Soriano BD, Buddhe S, Altman CA; EATAK Investigators. Etanercept With IVIg for Acute Kawasaki Disease: A Randomized Controlled Trial. Pediatrics. 2019 Jun;143(6):e20183675. doi: 10.1542/peds.2018-3675. Epub 2019 May 2. PMID 31048415
- [Result] Sagiv E, Slee A, Buffone A, Choueiter NF, Dahdah NS, Portman MA. Etanercept with IVIg for acute Kawasaki disease: a long-term follow-up on the EATAK trial. Cardiol Young. 2023 Apr;33(4):613-618. doi: 10.1017/S1047951122001470. Epub 2022 May 12. PMID 35545881

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo
  Placebo: Placebo 0.8 mg/kg subcutaneously (max 50 mg) given three times, once a week for three weeks starting at initial diagnosis.
Period: Overall Study
Arm/Group | Arm 1 -Etanercept | Placebo
Started | 103 | 102
Completed | 98 | 99
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: Kawasaki Disease Patients enrolled according to protocol who receive intravenous gamma-globulin as primary treatment.
Groups:
- Arm-2 Placebo: Placebo
  Placebo: Placebo 0.8 mg/kg subcutaneously (max 50 mg) given three times, once a week for three weeks starting at initial diagnosis.
- Total: Total of all reporting groups
Arm/Group | Arm 1 -Etanercept | Arm-2 Placebo | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100 | 101 | 201
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.77 (2.67) | 3.66 (2.75) | 3.70 (2.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 40 | 74
  Male | 66 | 61 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 17 | 36
  Not Hispanic or Latino | 81 | 84 | 165
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 14 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 54 | 60 | 114
  More than one race | 18 | 18 | 36
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Canada | 16 | 16 | 32
  United States | 84 | 85 | 169
KD Patients treated with IVIG [Count of Participants; unit: Participants] | 100 | 101 | 201

OUTCOME MEASURES:

1. Primary Outcome: IVIG Refractory
Description: The primary outcome is the proportion of subjects who become refractory to IVIG. Subjects requiring 1 dose of IVIG are classified as responders and subjects requiring more than 1 dose are classified as IVIG refractory.
Time Frame: 42 days after initial dose
Population: All patients receiving study drug
Measure: Count of Participants; unit: Participants
Groups:
- ARM 2 Placebo: Placebo
  Placebo: Placebo 0.8 mg/kg subcutaneously (max 50 mg) given three times, once a week for three weeks starting at initial diagnosis.
Arm/Group | Arm 1 -Etanercept | ARM 2 Placebo
Number analyzed (Participants) | 100 | 101
Participants | 13 | 22
Statistical Analysis 1: Comparison: Arm 1 -Etanercept vs ARM 2 Placebo; Test type: Superiority; p = .10, Chi-squared

2. Secondary Outcome: Determine if Etanercept Treatment Alters the Rate of Coronary Artery Dilation and Disease (CAD) at 2 and 6 Weeks After Treatment in Patients With Dilated Coro
Description: The primary echocardiographic outcome will be the proportion of subjects with improvement defined as (20% change in coronary artery) from the worst findings during the acute study period (scheduled visits from admission to visit 4, including any unscheduled visits) to the primary study outcome time-point at visit 5 (visit 5). This calculation will be based on changes in absolute values and not z-scores as initially planned. Groups will be compared using a logistic model including a binary term for age < versus > 1 year. Two aspects of the echo findings will be considered:
  * Maximum aneurysm size and
  * Maximum measurements for left main coronary artery (LMCA), left anterior descending artery (LAD) and right coronary artery (RCA).
  * Change in diameter of each coronary artery will be determined at standard measurement location or aneurysm with the latter taking precedent.
Time Frame: 42 days after initial dose
Population: All patients receiving study drug with coronary measures improved
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 -Etanercept | ARM 2 Placebo
Number analyzed (Participants) | 100 | 101
Participants | 56 | 53
Statistical Analysis 1: Comparison: Arm 1 -Etanercept vs ARM 2 Placebo; We applied a Generalized Estimating Equation (GEE) model to determine z score change values (see Protocol page 36 in Supplement); Test type: Superiority; p = 0.86, Regression, Cox

3. Other Pre Specified Outcome: Change in Coronary Artery Dimension by z Score Compared With General Estimating Equation
Description: Overall change in coronary z score over time determined using General Estimating Equation in patients from baseline within patients. No change or improved defined by 20% change in z score.
  A Z score normalized for body surface area represents how much larger (or smaller) a measured coronary artery internal diameter by echocardiography is compared to the average coronary artery diameter for a child of the same size (body surface area includes both height and weight). There is no minimum or maximum value. Z score above 2.0 is at least 2 standard deviations above mean for population and is considered abnormal. A decrease in z score is favorable.
Time Frame: 6 weeks
Population: Includes patients categorized by baseline coronary artery dilation (echocardiography) with stable or improved coronary artery z score
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Arm 1 -Etanercept | ARM 2 Placebo
Number analyzed (Participants) | 98 | 99
units on a scale | -0.4 (.122) | -0.10 (0.159)
Statistical Analysis 1: Comparison: Arm 1 -Etanercept vs ARM 2 Placebo; General Estimating Equation; Test type: Superiority; p = .83, GEE
Statistical Analysis 2: Comparison: Arm 1 -Etanercept vs ARM 2 Placebo; We analyzed change from baseline for both etanercept and placebo. LS mean change J(standard error) reported; Test type: Other — Generallzed Estimating Equation was used for z-score change within groups compared to baseline; p = 0.1279, GEE; General Estimating Equation

4. Other Pre Specified Outcome: Overall Change in z Score Over Time in Patients With Dilated Coronary Artery at Baseline Within Patients.
Description: Overall change in z score over time determined using General Estimating Equation in patients with dilated coronary artery at baseline within patients. Overall change in coronary z score over time determined using General Estimating Equation in patients from baseline within patients. A Z score normalized for body surface area represents how much larger (or smaller) a measured coronary artery internal diameter by echocardiography is compared to the average coronary artery diameter for a child of the same size (body surface area includes both height and weight). There is no minimum or maximum value. Z score above 2.0 is at least 2 standard deviations above mean for population and is considered abnormal. A decrease in z score is favorable.
Time Frame: 6 weeks
Population: KD patients with dilated coronary arteries at baseline (improved or stable)
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arm 1 -Etanercept | ARM 2 Placebo
Number analyzed (Participants) | 24 | 22
score on a scale | -081 (0.39) | 0.4 (0.81)
Statistical Analysis 1: Comparison: Arm 1 -Etanercept; General Estimating Equation; Test type: Other — General Estimating Equation for 3 coronary arteries; p = 0.03, GEE; Generalize estimating equation for 3 coronary arteries evaluated in each patient by echocardiography
Statistical Analysis 2: Comparison: ARM 2 Placebo; GEE performed to compare with change in coronary z score from baseline; Test type: Other — see above; p = 0.619, GEE

ADVERSE EVENTS:
Time Frame: 42 days
Description: Does not differ from clinicaltrials.gov
Groups:
- Arm -2 Placebo: Placebo
  Placebo: Placebo 0.8 mg/kg subcutaneously (max 50 mg) given three times, once a week for three weeks starting at initial diagnosis.
Arm/Group | Arm 1 -Etanercept | Arm -2 Placebo
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/102
Serious Adverse Events (participants affected / at risk) | 9/99 | 10/102
Other Adverse Events (participants affected / at risk) | 10/99 | 12/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 -Etanercept (N=99) | Arm -2 Placebo (N=102)
Hospital readmission for retreatment (Immune system disorders) | 7 (7) | 10 (10) — Hospital readmission for retreatment of KD
Infection (Infections and infestations) | 2 | 0 — Infection
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 -Etanercept (N=99) | Arm -2 Placebo (N=102)
Skin Rash (Skin and subcutaneous tissue disorders) | 10 (10) | 12 (12) — RASH

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-07-06): https://cdn.clinicaltrials.gov/large-docs/89/NCT00841789/Prot_SAP_000.pdf